CLINICAL TRIAL: NCT02013661
Title: Clinical Evaluation of Four Types of Suture in Periodontal Surgery
Brief Title: Clinical Evaluation of Sutures in Periodontal Surgery
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Almudena Tasende Pereiro, DDS, Ms., Universitat Internacional de Catalunya
Other Study IDs: C-12-ASA-10
Record Dates: First submitted 2013-11-27; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Periodontal Debridement
Keywords: periodontal debridement; sutures; tissue reaction

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suture in Periodontal resective surgery: Four types of suture including silk, polypropylene, PGA, and PTFE
  Interventions: Procedure: Periodontal resective surgery

INTERVENTIONS:
Procedure: Periodontal resective surgery — surgical periodontal debridement is performed after periodontal phase I

SUMMARY:
The aims of this study were to evaluate and compare tissue erythema, edema and knot loosening among four types of suture one week after periodontal surgery.

DETAILED DESCRIPTION:
Forty patients participated in this prospective, randomized, double-blind clinical trial. Vertical mattress sutures were used following resective periodontal surgery performed by one operator. Four suture materials were selected for evaluation: 5-0 silk; 5-0 polypropylene; 5-0 polyglycolic acid (PGA), and 4-0 polytetrafluoroethylene (PTFE). Seven days after the surgical procedure, the surgeon assessed suture loosening and removed the sutures. A blind researcher clinically evaluated erythema and edema.

ELIGIBILITY:
Inclusion Criteria:

* Qualification for the study was based on the need for resective periodontal surgery (apically positioned flap and osseous recontouring) at four or more consecutive interproximal sites per quadrant

Exclusion Criteria:

* systemic diseases, such as diabetes, chronic obstructive pulmonary disease, or an immunologic disease that would affect wound healing; allergies to prescribed medication; and/or current pregnancy or breast feeding were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients treated at the CUO (dental clinic at the Universitat Internacional de Catalunya) that are prescribed for periodontal resective surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
presence or absence of Suture loosening | seven days after surgery
  Seven days after the surgical procedure, the surgeon assessed suture loosening; recording loose or not Loose

SECONDARY OUTCOMES:
presence and level of erythema and edema. | seven days after surgery
  Seven days after the surgical procedure a blind researcher clinically evaluated erythema and edema. Adding a score related to a gingival index

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, DDS, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, San Cugat Del Valles, Barcelona, Spain